CLINICAL TRIAL: NCT04166851
Title: Using Open Contest and Neuro-influence Experiment to Develop and Evaluate PrEP Promotion Messages for High Risk Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00008650
Record Dates: First submitted 2019-10-23; First posted 2019-11-18 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS
Keywords: Pre-exposure prophylaxis; Health Promotion; HIV/AIDS primary prevention; men who have sex with men; Neuroimaging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open contest messages (Experimental): Participants will view the top PrEP-promotion messages developed via an open contest.
  Interventions: Behavioral: PrEP campaign messages developed via open contest
- Social marketing messages (Active Comparator): Participants will view the PrEP-promotion messages developed via social marketing.
  Interventions: Behavioral: PrEP campaign messages developed via social marketing approach

INTERVENTIONS:
Behavioral: PrEP campaign messages developed via open contest — PrEP campaign messages will be developed via an open contest in Baltimore.
  Arms: Open contest messages
Behavioral: PrEP campaign messages developed via social marketing approach — PrEP campaign messages developed with a traditional social marketing approach.
  Arms: Social marketing messages

SUMMARY:
The aim of this study is to examine the utility of neuroimaging technique to evaluate pre-exposure prophylaxis (PrEP) promotion messages for men who have sex with men (MSM) at risk of HIV in Baltimore.

DETAILED DESCRIPTION:
This study will examine the utility of neuroimaging technique to evaluate PrEP promotion messages for MSM at risk of HIV in Baltimore. The investigators hypothesize that participants viewing top messages developed via open contests will show higher brain activation in the Medial Prefrontal Cortex (MPFC) regions than those viewing messages developed by a social marketing approach. The investigators further hypothesize brain activation in the MPFC regions is significantly more correlated with PrEP behavioral intention, initiation, and action than self-reported message effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Biological male sex at birth
* Sexually active with men in the past 6 months
* Never taken PrEP
* HIV negative
* Reside in Baltimore City or surrounding counties
* Meet one of the criteria for being an appropriate PrEP candidate (i.e. in a relationship with a partner not known to be HIV-negative; are in a nonmonogamous relationship; have had any condomless anal sex with a casual male partner regardless of status in the prior 6 months; or had a positive sexual transmitted infection (STI) diagnosis within the prior 6 months).

Exclusion Criteria:

- Participated in open contest

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cui Yang, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Contest Messages | Social Marketing Messages
Started | 14 | 9
Completed | 14 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Contest Messages | Social Marketing Messages | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 34 [23 to 65] | 32 [24 to 56] | 33 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 9 | 23
Interntion to use PrEP [Mean (Standard Deviation); unit: units on a scale] — Suppose that PrEP is at least 90% effective in preventing HIV when taken as prescribed. How likely would you plan to take PrEP if it were available for free?
  1. Extremely unlikely
  2. Somewhat unlikely
  3. Somewhat likely
  4. Extremely likely
  Mean of participant choice is reported Population: Some participants didn't answer due to skip pattern in survey
  units on a scale
    number analyzed (Participants) | 12 | 5 | 17
    (all) | 3 (1.20) | 3.6 (0.55) | 3.18 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Change of Willingness to Take PrEP
Description: Questions on willingness to take PrEP. Participants will be asked, "Suppose that PrEP is at least 90% effective in preventing HIV when taken daily. How likely would you be to take PrEP if it were available for free?" with responses ranging from "Extremely unlikely-1," "Somewhat unlikely-2," "Somewhat likely-3," "Extremely likely-4." The mean of the changes between baseline and after participants reviewed the messages was calculated.
Time Frame: baseline, 30 days post baseline
Population: Participants who completed the follow-up survey are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Contest Messages | Social Marketing Messages
Number analyzed (Participants) | 5 | 2
units on a scale | 0 (0) | 0.5 (0.71)

ADVERSE EVENTS:
Description: Adverse Events Were Not Collected
Arm/Group | Open Contest Messages | Social Marketing Messages
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT04166851/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04166851/ICF_001.pdf